CLINICAL TRIAL: NCT00942669
Title: A Prospective, Single Center, Open, Equivalence, Two Phase Study Comparing the Sleep Strip OTC™ Accuracy in Screening for Sleep Apnea Syndrome Against the Reference Method, an In-lab Full Night Polysomnographic (PSG) Study.
Brief Title: Comparing the Sleep Strip OTC™ Accuracy in Screening for Sleep Apnea Syndrome Against the Reference Method, an In-lab Full Night Polysomnographic (PSG)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Scientific Laboratory Products, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SS-OTC-346 CTIL
Record Dates: First submitted 2009-07-11; First posted 2009-07-21 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Sleep Apnea Syndrome
Keywords: Sleep Apnea Syndrome; SAS; SleepStrip OTC
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SleepStrip OTC(TM) (Experimental): Participants will receive the SleepStrip OTC(TM) for a night (or two) test at home, before or after undergoing an independent PSG test at the Sleep lab. The reading of both methods will be analyzed.
  Interventions: Device: SleepStrip OTC(TM)

INTERVENTIONS:
Device: SleepStrip OTC(TM) — self contained SAS screening device
  Other Names: SleepStrip OTC; SAS; Sleep Apnea; PSG

SUMMARY:
The primary purpose of this study is to demonstrate the equivalence of the new Sleep Strip OTC(TM) compared to the reference method of an in-lab, attended full-night polysomnographic (PSG) study.

DETAILED DESCRIPTION:
A prospective, single center two phase study to evaluate the validity and the predictability of the SleepStrip OTCTM in screening for SAS, as compared to the reference method, an in-lab, full night, attended Polysomnographic (PSG) Study.

The study will consist of two phases:

I: Optimization Phase:will be performed at the Clinic; 20 participants will be enrolled. Each participant will be connected simultaneously to the SleepStrip OTC(TM) and to the standard lab sensors and recorder. This phase is intended to allow SLP to optimize the analysis parameters for optimal performance and will be considered as a pilot phase.

II: Equivalence phase: At least 180 participants will be enrolled. All participants will receive the SleepStrip OTC(TM) for a night test at home, before or after undergoing an independent PSG test at the Sleep lab. Out of 180 participants, at least 26 participants will receive two SleepStrip OTC(TM) devices for two consecutive night tests at home. The remaining participants will receive one SleepStrip OTC(TM) for one night test.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female participants, 18 years of age or older at time of enrollment.
* Participants who present at the Technion Sleep Disorder Center for a PSG test, and who are willing comply with study procedures.
* Participants who are willing to sign a Written.

Exclusion Criteria:

* Participant has a clinically significant untreated chronic disease which may unable him/ her to participate in the study.
* Participant has facial hair or any other skin problem that may hinder proper application of the device on destined facial area.
* Participant is suffering from a respiratory-track infection or a runny nose at enrollment.
* Participant is unable to comprehend the purpose of the study as stated in the participant consent form.
* Participant is unable to comply with the technical requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Paired T-test or signed-rank test; McNemar's test; Sensitivity Analyses | The data will be analyzed after conclusion of tests of 200 home studies, no later than June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Giora Pillar, Prof., Principal Investigator — Technion Sleep Disorders Center, Rambam Medical Centaer, Israel
Locations (1):
- The Technion Sleep Disorders Center, Rambam Medical Center, Haifa, Israel